CLINICAL TRIAL: NCT00719576
Title: A Prospective, Randomized, Open-label, Parallel-group, Multi-center Study to Demonstrate the Superiority of MACI® Versus Arthroscopic Microfracture for the Treatment of Symptomatic Articular Cartilage Defects of the Femoral Condyle Including the Trochlea.
Brief Title: Superiority of MACI® Versus Microfracture Treatment in Patients With Symptomatic Articular Cartilage Defects in the Knee
Acronym: SUMMIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MACI00206; 2006-004817-16 (EudraCT Number)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Articular Cartilage Defect
Keywords: Cartilage legions; symptomatic focal cartilage defects; microfracture; MACI; autologous chondrocyte
MeSH Terms: conditions — Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MACI (Experimental): autologous cultured chondrocytes on porcine collagen membrane
  Interventions: Biological: autologous cultured chondrocytes on porcine collagen membrane
- Microfracture (Active Comparator): Microfracture
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Biological: autologous cultured chondrocytes on porcine collagen membrane — Implantation via mini-arthrotomy
  Other Names: MACI; matrix-applied characterized autologous cultured chondrocytes
  Arms: MACI
Procedure: Microfracture — Microfracture performed by arthroscopic surgery
  Arms: Microfracture

SUMMARY:
The objective of this trial is to demonstrate superior efficacy and safety of MACI compared with arthroscopic microfracture in the treatment of patients (aged 18 to 55 years) with symptomatic articular cartilage defects of the knee.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, parallel-group, multicenter study designed to investigate the outcome of MACI implant versus arthroscopic microfracture in the treatment of articular cartilage defects in the knee in patients between ages of 18 and 55 years.

All patients who meet the eligibility criteria and are considered suitable for inclusion will have a cartilage biopsy taken prior to randomization to study treatment. Eligible patients will then be randomized during the index arthroscopy procedure to receive either MACI implant or microfracture treatment.

Patients randomized to treatment with MACI implant will return within approximately 4 to 8 weeks of the index arthroscopy to undergo the chondrocyte implantation procedure via arthrotomy. Patients randomized to microfracture will undergo the procedure during the index arthroscopy.

Patients will be assessed post-arthroscopy and post-arthrotomy at intervals during 2 years follow-up. Evaluations include adverse events, functional and pain outcomes, arthroscopic and histologic evaluation and magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, single or multiple full-thickness cartilage defects of the knee with or without bone involvement

Exclusion Criteria:

* Known history of hypersensitivity to gentamicin, other aminoglycosides, or products of porcine or bovine origin
* Severe osteoarthritis of the knee
* Inflammatory arthritis, inflammatory joint disease, or uncorrected congenital blood coagulation disorders
* Prior knee surgery (within 6 months), excluding surgery to procure a biopsy or a concomitant procedure to prepare the knee for a MACI implant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (20):
- Czechia (3):
  - Urazova nemocnice v Brne, Brno
  - Fakultni Nemocnice Na Bulovce, Prague
  - Fakultni Nemocnice v Motole, Prague
- France (4):
  - Hopital d'instruction des armees Robert Picque, Bordeaux
  - Centre Hospitalier Lyon Sud, Lyon
  - Polyclinique Saint-Roch, Montpellier
  - Chirurgien Orthopediste et Traumatologue du Sport, Institut de I'Appareil Locomoteur Nollet, Paris
- Netherlands (3):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Elisabeth Ziekenhuis, Tilburg
  - UMC Utrecht, Utrecht
- St Olavs Hospital, Trondheim, Norway
- Poland (4):
  - Szpital Uniwersytecki, Bydgoszcz
  - Regional Hospital of Traumatologic Surgery, Piekary Śląskie
  - Center for Sports Medicine CMS, Warsaw
  - Medical Academy Warsaw, Warsaw
- Sweden (2):
  - Kungsbacka Hospital, Kungsbacka
  - Capio Artro Clinic AB, Stockholm
- United Kingdom (3):
  - The South West London Elective Orthopaedic Centre (SWLEOC), Epsom
  - Nuffield Dept. of Orthopaedic Surgery, University of Oxford, Oxford
  - Spire Cheshire Hospital, Warrington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saris D, Price A, Widuchowski W, Bertrand-Marchand M, Caron J, Drogset JO, Emans P, Podskubka A, Tsuchida A, Kili S, Levine D, Brittberg M; SUMMIT study group. Matrix-Applied Characterized Autologous Cultured Chondrocytes Versus Microfracture: Two-Year Follow-up of a Prospective Randomized Trial. Am J Sports Med. 2014 Jun;42(6):1384-94. doi: 10.1177/0363546514528093. Epub 2014 Apr 8. PMID 24714783

RESULTS

PARTICIPANT FLOW:
Groups:
- Microfracture: Microfracture
  Microfracture: Microfracture
Period: Overall Study
Arm/Group | MACI | Microfracture
Started | 72 | 72
Completed | 70 | 67
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MACI | Microfracture | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (9.16) | 32.9 (8.78) | 33.8 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 45 | 48 | 93
Region of Enrollment [Number; unit: participants]
  Czech Republic | 13 | 11 | 24
  Netherlands | 28 | 30 | 58
  Sweden | 1 | 1 | 2
  Norway | 3 | 3 | 6
  Poland | 14 | 14 | 28
  United Kingdom | 4 | 4 | 8
  France | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 104 for the Participant's Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain and Function (Sports and Recreational Activities) Scores.
Description: The KOOS is a validated knee-specific instrument developed to assess the patients' opinion of their knee and associated problems. KOOS consists of 5 subscales: Pain, Function in sports and recreational activities, other Symptoms, Function in activities of daily living (ADL), and knee related Quality of life (QOL). A 5-point Likert scale was used to record the response to each item ranging from 0 (no problems) to 4 (extreme problems). Within each subscale, items were added up and normalized to a value between 0 (extreme problems) and 100 (no problems). Subscales are not combined to calculate a total score.
Time Frame: Baseline and Week 104
Population: All randomized patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 72 | 72
units on a scale
  Change from Baseline KOOS Pain | 45.45 (21.08) | 35.23 (23.91)
  Change from Baseline KOOS Function | 46.04 (28.35) | 35.83 (31.63)
Statistical Analysis 1: Comparison: MACI vs Microfracture; The changes from Baseline to Week 104 in KOOS Pain and Function (SRA) scores (co-primary efficacy parameter) were analyzed with a multivariate analysis of variance (MANOVA) model, with the last observation carried forward (LOCF) method for handling missing data. Terms included in the model are treatment and center as class variables and baseline KOOS pain and Function (SRA) as continuous covariates; Test type: Superiority — The Wilks lambda test statistic and associated single P value from the MANOVA model were used to test the statistical significance of the difference in the co-primary endpoint between MACI and microfracture; p = 0.001, MANOVA

2. Secondary Outcome: Histological Evaluation of Structural Repair of Evaluable Biopsies Harvested From the Core of the Index Lesion During Arthroscopy at Week 104
Description: The mean microscopic International Cartilage Repair Society (ICRS) II overall assessment score was used to assess the histology efficacy endpoint.
  Scoring of the cartilage repair biopsies was completed using the ICRS II histology scoring system (Mainil-Varlet, 2010, Am J Sports Med) by 2 independent pathologists blinded to the patient's assigned study treatment. This scoring system includes 14 parameters, comprising an overall assessment score reported here, as well as 13 other items related to chondrocyte phenotype, tissue structure, and other factors, each scored on a scale from 0 to 100 representing poor to good quality cartilage.
Time Frame: Week 104
Population: includes all subjects with histology follow-up data
Measure: Least Squares Mean (Full Range); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 60 | 56
units on a scale | 63.8 [0 to 95] | 62.3 [7 to 97]
Statistical Analysis 1: Comparison: MACI vs Microfracture; Test type: Superiority or Other; p = .717, ANOVA — Differences between groups were tested using analysis of variance; ANOVA with terms for treatment and center

3. Secondary Outcome: Assessment of Defect Fill by Magnetic Resonance Imaging (MRI)
Description: Number of participants with MRI degree of defect fill > 50%. Evaluation of MRI data was performed by independent central review blinded to the participant's treatment.
  Appropriate MRI sequences were used to image cartilage repair tissue.
Time Frame: Week 104
Population: Number of participants with MRI data at Week 104
Measure: Count of Participants; unit: Participants
Groups:
- Microfracture: Microfracture: Microfracture
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 70 | 69
Participants | 58 | 53
Statistical Analysis 1: Comparison: MACI vs Microfracture; Differences between groups were tested by the Cochran-Mantel-Haenszel row mean score chi-squared test for defect fill; Test type: Superiority; p = .920, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Row Mean Score Chi-Square

4. Secondary Outcome: Response Rate Based on KOOS Pain and Function (Sports and Recreational Activities) Scores at Week 104.
Description: A responder is defined as a participant with at least a 10-point improvement in both the KOOS Pain and Function (Sports and Recreational activities) scores from Baseline
Time Frame: Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 72 | 72
Participants | 63 | 49
Statistical Analysis 1: Comparison: MACI vs Microfracture; Differences between groups were tested by the Cochran-Mantel-Haenszel chi-squared test stratified by center for responders; Test type: Superiority; p = 0.016, Cochran-Mantel-Haenszel — KOOS Response Rate: a participant is regarded as a responder for KOOS if a 10-point improvement in both KOOS Pain and Function (SRA) scores was achieved with respect to Baseline. Otherwise, the patient is regarded as a nonresponder; p-value was calculated for response categories 'Responded' and 'Not responded' using a Cochran-Mantel-Haenszel χ2 Test stratified by Center

5. Secondary Outcome: Treatment Failure
Description: The planned analyses concerning time to treatment failure were not conducted due to the small number of per protocol treatment failure cases. As such, the number of participants with treatment failure is being reported.
  Patients were considered as a treatment failure if all of the following 5 criteria were met:
  1. Patient's global assessment of their knee joint compared to Baseline was the same or worse
  2. Physician's global assessment of the patient's knee joint compared to Baseline was the same, worse, or significantly worse.
  3. Percent improvement from Baseline in KOOS Pain score was less than 10%.
  4. Physician diagnostic evaluation of failure excluded etiologies (eg, meniscal tear) other than failed treatment of the index lesion.
  5. The physician decided that surgical re-treatment of the index lesion(s) was required that involved either extensive debridement for lesion expansion, violation of the subchondral bone, or autologous cultured chondrocyte implantation.
Time Frame: Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 72 | 72
Participants | 0 | 2

6. Secondary Outcome: Change From Baseline at Week 104 in the Remaining 3 Subscales of the KOOS Instrument (Activities of Daily Living, Knee-related Quality of Life, and Other Symptoms)
Description: The KOOS is a validated knee-specific instrument developed to assess the patients' opinion of their knee and associated problems. KOOS consists of 5 subscales: Pain, Function in sports and recreational activities, other Symptoms, Function in activities of daily living (ADL), and knee related Quality of life (QOL). A 5-point Likert scale was used to record the response to each item ranging from 0 (no problems) to 4 (extreme problems). Within each subscale, items were added up and normalized to a value between 0 (extreme problems) and 100 (no problems).
Time Frame: Baseline and Week 104
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 72 | 72
units on a scale
  Change from Baseline in Activities of Daily Living | 43.70 (24.52) | 32.76 (26.78)
  Change from Baseline in KOOS Quality of Life | 37.41 (27.24) | 29.93 (28.11)
  Change from Baseline in KOOS Other Symptoms | 35.47 (20.83) | 27.31 (24.59)
Statistical Analysis 1: Comparison: MACI vs Microfracture; Analysis of covariance was conducted with treatment and center as fixed effects and Baseline subscale as covariate, conducted at α = 0.05 level of significance. Last observation carried forward was used for missing data imputation; Test type: Superiority; p < 0.001, ANCOVA — KOOS activities of daily living p-value <0.001
Statistical Analysis 2: Comparison: MACI vs Microfracture; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.029, ANCOVA — KOOS knee-related quality of life p-value 0.029
Statistical Analysis 3: Comparison: MACI vs Microfracture; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — KOOS other symptoms p-value <0.001

7. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Time Frame: Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 72 | 72
Participants | 55 | 60

ADVERSE EVENTS:
Time Frame: Week 104
Arm/Group | MACI | Microfracture
Serious Adverse Events (participants affected / at risk) | 11/72 | 19/72
Other Adverse Events (participants affected / at risk) | 55/72 | 58/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MACI (N=72) | Microfracture (N=72)
Arrhythmia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 1
Treatment failure (General disorders) | 1 | 4
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 2 | 6
Graft delamination (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MACI (N=72) | Microfracture (N=72)
Pyrexia (General disorders) | 4 | 2
Influenza (Infections and infestations) | 4 | 5
Nasopharyngitis (Infections and infestations) | 10 | 7
Procedural pain (Injury, poisoning and procedural complications) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Joint effusion (Musculoskeletal and connective tissue disorders) | 5 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 7 | 4
Ligament sprain (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 13 | 21
Abdominal Pain (Gastrointestinal disorders) | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 46

LIMITATIONS AND CAVEATS:
Because clinical trials are conducted under widely varying conditions, adverse event rates observed in clinical trials cannot be directly compared to rates in the clinical trials of another product and may not reflect the rates observed in practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days